CLINICAL TRIAL: NCT02281539
Title: Myoelectrically Controlled Augmented Reality and Gaming for the Treatment of Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrum (Industry)
Collaborators: Sahlgrenska University Hospital (Other); Region Örebro County (Other); Bräcke diakoni Rehabcenter Sfären (Unknown); University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLP-004664
Record Dates: First submitted 2014-10-12; First posted 2014-11-03 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Phantom Limb Pain
Keywords: Phantom Limb Pain; Augmented Reality; Myoelectric control; Virtual reality; electromyography; pattern recognition; neurorehabilitation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment using myoelectric signals (Experimental): Virtual- and augmented reality, are controlled by the patient's phantom limb using muscle (myoelectric) signals from the stump. The patient learns to reactivate areas in the brain related to motor control of the missing limb. The medical device is non-invasive and based on surface electromyography
  Interventions: Device: Neuromotus

INTERVENTIONS:
Device: Neuromotus

SUMMARY:
The goal of the clinical investigation is to reduce phantom limb pain (PLP), painful condition affecting 70% of amputees, so as to improve these patients' quality of life.

DETAILED DESCRIPTION:
The goal of the clinical investigation is to reduce phantom limb pain (PLP), a painful condition affecting 70% of amputees, so as to improve these patients' quality of life. Traditionally, mirror box therapy and other tools based on the same concept, have been used to alleviate pain, but their efficacy varies greatly. This project targets amputees for whom other PLP treatments have failed. Various virtual environments, including virtual/augmented reality, are controlled by the patient's phantom limb using muscle (myoelectric) signals from the stump. The patient learns to reactivates areas in the brain related to motor control of the missing limb.

The medical device is non-invasive and based on surface electromyography, a standard and widely used clinical and research tool. The surface electrodes are a standard disposable electrodes widely used in clinics and hospitals for EMG and/or ECG.

* Myoelectric amplifiers (battery operated and isolated from the power grid)
* Data acquisition electronics
* Personal computer
* Standard webcam
* Myoelectric pattern recognition (MPR) software
* Virtual Reality (VR)
* Augmented Reality (AR)
* Computer game

The clinical investigation period consists of 12 sessions per patient including 3 short follow-up assessments. Length of the session: 1.5 hours (the first sessions can take longer time due to learning/familiarization). The centers participating in this study can choose between the following treatment administrations:

* 2 times per week (advised)
* 1 time per week
* Daily (5 times per week)

ELIGIBILITY:
Inclusion Criteria:

* Amputee patients older than 18 years.
* The patient has signed a written informed consent.
* Patients must have been treated with at least one of the following therapies:

  1. Conventional mirror training
  2. Transcutaneous electrical stimulation (TENS)
  3. Acupuncture
  4. Self-hypnosis
  5. Drug-based
* The last session of previous therapies (1 and 2) must be at least 1 month before beginning the treatment here proposed.
* In the case of drug-based treatments (5), the patient must report no PLP reduction for at least 1 month under the drug-based treatment and no variations on the medicaments dose. Any pain reduction potentially attributed to the drug-based treatment must be at least 3 months old.
* At least a portion of biceps and triceps muscles must be present.

Exclusion Criteria:

* Patient must not have a significant cognitive impairment that prevents them from following instructions.
* Upper limb amputees excluding shoulder disarticulation.
* Obese patient will not be automatically excluded, however, an evaluation in the system is required to analyse if sufficient electromyography signals can be recorded.
* Stump pain over 2 VAS of pain.
* Participating in any other clinical study that could interfere with the result in the ongoing study.
* Condition associated with risk of poor protocol compliance.
* Any other condition or symptoms preventing the patient from entering the study, according to the investigator´s judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Measuring the portion of patients that had a reduction of PLP according to the calculated weighted pain distribution (WPD) | 12 treatment sessions (up to 12 weeks) + follow up (6months). Time frame will be total of 9 months.
  Each patient is asked to estimate the time spent in a given level of pain (as by VAS). The WPD is the sum of the portion of time multiplied with the pain level (0 to 5). This can also be explained as weighted mean calculation. The time with a given level of pain can be estimated in minutes/hours and extrapolated to its corresponding portion from the total time. Phantom Limb pain, which is a chronic pain, is difficult to describe can not be assesst in a single point in time. That is why patients are asked to fill in the amount of time they spend in each level of pain.

SECONDARY OUTCOMES:
Descriptive analysis on the effect of the proposed treatment on quality of life, disability at the activity and participation levels.(DASH/COPM/EQ-5D) | 12 treatment sessions (up to 12 weeks) + follow up (6months). Time frame will be total of 9 months.
  Questionnaires are answered before the first treatment and after the last treatment. Patients will also answer the questionnaires for a follow-up.
Measure the portion of patients that had a reduction of PLP with the use of visual analog scale and reduction on the "pain rating index". | 12 treatment sessions (up to 12 weeks) + follow up (6months). Time frame will be total of 9 months.
  For the Pain Rating Index (PRI), each selected word is scored from 0 (none) to 5 (Excruciating pain). The total Pain Rating Index score is obtained by summing the item scores and higher score indicates worse pain.
Descriptive analysis on the effect of the proposed treatment in medicaments intake | 12 treatment sessions (up to 12 weeks) + follow up (6months). Time frame will be total of 9 months.
  questionnaires compared
Patients having the same treatment administration will be classified in subgroups and their results compared. | 12 treatment sessions (up to 12 weeks) + follow up (6months). Time frame will be total of 9 months.
  questionnaires compared

CONTACTS AND LOCATIONS:
Overall Officials: Rickard Brånemark, MD MSC, PhD, Study Chair — Integrum AB; Kerstin Caine-Winterberger, OT, Principal Investigator — Rehabilitation Center for Upper Limb Prosthetics, Sahlgrenska University Hospital
Locations (1):
- Rehabilitation Center for Upper Limb Prosthetics, Gothenburg, Sweden

REFERENCES:
- [Result] Ortiz-Catalan M, Sander N, Kristoffersen MB, Hakansson B, Branemark R. Treatment of phantom limb pain (PLP) based on augmented reality and gaming controlled by myoelectric pattern recognition: a case study of a chronic PLP patient. Front Neurosci. 2014 Feb 25;8:24. doi: 10.3389/fnins.2014.00024. eCollection 2014. PMID 24616655
- [Derived] Ortiz-Catalan M, Guethmundsdottir RA, Kristoffersen MB, Zepeda-Echavarria A, Caine-Winterberger K, Kulbacka-Ortiz K, Widehammar C, Eriksson K, Stockselius A, Ragno C, Pihlar Z, Burger H, Hermansson L. Phantom motor execution facilitated by machine learning and augmented reality as treatment for phantom limb pain: a single group, clinical trial in patients with chronic intractable phantom limb pain. Lancet. 2016 Dec 10;388(10062):2885-2894. doi: 10.1016/S0140-6736(16)31598-7. Epub 2016 Dec 2. PMID 27916234